CLINICAL TRIAL: NCT03986853
Title: Exploration of Angiogenesis in Decompensated Developmental Venous Abnormalities
Acronym: Explor-AVD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Patient with rare disease
Sponsor: Hopital Foch (Other)
Collaborators: Collège de France (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2017007-F
Record Dates: First submitted 2019-06-13; First posted 2019-06-14 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Developmental Venous Anomaly
MeSH Terms: conditions — Central Nervous System Venous Angioma | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blood sample (Experimental): Blood sampling Under general anesthesia
  Interventions: Procedure: Blood sampling

INTERVENTIONS:
Procedure: Blood sampling — Blood sampling under general anesthesia

SUMMARY:
The purpose of our study is to demonstrate by blood samples in situ in the vascular lesion (performed during any cerebral catheterization for an embolization of arteriovenous malformation) the existence of angiogenic growth factors and inflammatory factors that would confirm the decompensation of venous ischemia.

ELIGIBILITY:
Main Inclusion Criteria:

* Presenting a DVA requiring hyperselective catheterization
* Having sign an informed consent form

Exclusion Criteria:

* Presenting a contraindication to the realization of hyperselective cathterism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-01-11 (Actual); Primary Completion 2021-01-11 (Actual); Study Completion 2021-01-11 (Actual)

PRIMARY OUTCOMES:
Assessment of angiogenic and inflammatory growth factors | 1 day
  The 1st factor studied is VEGF-A
Assessment of angiogenic and inflammatory growth factors | 1 day
  The 2nd factor studied is VEGF-A
Assessment of angiogenic and inflammatory growth factors | 1 day
  The 3rd factor studied is angiopoitin-2
Assessment of angiogenic and inflammatory growth factors | 1 day
  The 4th factor studied is PDGF
Assessment of angiogenic and inflammatory growth factors | 1 day
  The 5th factor studied is angiopoietin-like 4

CONTACTS AND LOCATIONS:
Overall Officials: Georges Rodesch, Principal Investigator — Hôpital Foch
Locations (1):
- Hôpital Foch, Suresnes, France